CLINICAL TRIAL: NCT01907048
Title: Xarelto (Rivaroxaban) Risk Minimisation Plan Evaluation: Patient and Physician Knowledge of Key Safety Messages
Brief Title: Patient and Physician Knowledge of Key Safety Messages
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry); RTI Health Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: 16167; XA1202 (Other: Company Internal)
Record Dates: First submitted 2013-06-12; First posted 2013-07-24 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Anticoagulation
Keywords: Survey; Effectiveness of risk minimization measures; Rivaroxaban; Anticoagulants
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Survey to measure physician awareness and understanding of the key messages in the prescriber guide.
  Interventions: Behavioral: Rivaroxaban (Xarelto, BAY59-7939)
- Group 2: Survey to measure patient awareness and understanding of the key messages in the patient card.
  Interventions: Behavioral: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Behavioral: Rivaroxaban (Xarelto, BAY59-7939) — Survey to measure physician awareness and understanding of the key messages in the prescriber guide.
  Groups: Group 1
Behavioral: Rivaroxaban (Xarelto, BAY59-7939) — Survey to measure patient awareness and understanding of the key messages in the patient card.
  Groups: Group 2

SUMMARY:
This cross-sectional epidemiologic study measured physician and patient awareness and understanding of the key messages in the Xarelto prescriber guide and Xarelto patient alert card.

ELIGIBILITY:
- Inclusion criteria:

Physician eligibility:

* Prescription of rivaroxaban in the past 6 months for adult patients for the Prevention of stroke and systemic embolism with non-valvular atrial fibrillation (SPAF) or Treatment of deep venous thrombosis (DVT) and prevention of recurrent DVT and pulmonary embolism (PE) following an acute DVT.

Patient eligibility:

* Use of rivaroxaban for SPAF or DVT within the previous 3 months; aged 18 years and above; able to understand and complete the consent form and patient questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians of various specialties; patients treated in primary care and specilized clinical practices.
Sampling Method: Non-Probability Sample
Enrollment: 2227 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Knowledge and understanding among physicians regarding key safety information contained in the prescriber guide assessed by web-based questionnaire | Up to 18 months
Knowledge and understanding of patients regarding the key safety information contained in the patient alert card assessed by paper-based questionnaire | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Multiple Locations, France
- Multiple Locations, Germany
- Multiple Locations, Spain
- Multiple Locations, United Kingdom

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/